CLINICAL TRIAL: NCT03039907
Title: A Critical Assessment of the Factors That Promote or Limit the Return to Recreational, Work, and Physical Fitness Activities After Primary Total Knee Arthroplasty
Brief Title: Return to Physical Activities After Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cincinnati Sportsmedicine Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Sue Barber-Westin, Director Clinical Studies, Cincinnati Sportsmedicine Research and Education Foundation
Other Study IDs: TKAUnder65-001
Record Dates: First submitted 2016-04-11; First posted 2017-02-01 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Knee; Replacement
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Total knee arthroplasty

SUMMARY:
The main purpose of this study is to examine the factors that allow patients that undergo total knee arthroplasty to return to recreational sports and/or work activities, and to achieve recommended physical activity levels.

DETAILED DESCRIPTION:
There are three purposes of this study. The first purpose is to examine the factors that allow patients that underwent total knee arthroplasty with the Journey II to return to recreational sports and/or work activities, and to achieve recommended physical activity levels (defined by the American Heart Association and the American College of Sports Medicine).

The second purpose is to examine the factors that limit the ability of patients to resume sports, work, and physical fitness training, including comorbidities, general health, complications, and other factors.

The third purpose is to use advanced sports medicine rehabilitation principles that involve staged progressive protocols to safely prepare patients for sports, work, and physical fitness training. Objective measurements of muscle strength, endurance, balance, and neuromuscular control will be used to determine when patients may be cleared to participate in these activities.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 65 years of age or younger.
* Patient indicates before surgery the desire to return to recreational (sports) and/or work activities postoperatively
* Patient provides informed consent.
* Patient complies with postoperative rehabilitation program.

Exclusion Criteria:

* Patient did not desire to return to recreational and/or work activities after TKA
* History of alcohol or drug abuse within 3 years of the operation.
* Disabling or widespread osteoarthritis or other joint disease in any other joint.
* Presence of a significant connective tissue disease, autoimmune disease, HIV-positive, or immune deficiency syndrome.
* Any other contraindications that in the opinion of the principal investigator would interfere with the conduct of the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 65 years of age and younger who undergo total knee arthroplasty who desire to return to recreational (sports) and/or work activities postoperatively.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01-23 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of Number of Participants That Return to Recreational and Fitness Activities | 2 years postoperatively
  Participants will complete a questionnaire that determines the type of physical activities they routinely participate in (for instance, swimming, bicycling, hiking, golf). Patients will also complete two questions regarding their general fitness level in accordance with current standards of the American Heart Association. These questions are contained in the study patient registry.

SECONDARY OUTCOMES:
Assessment of Effect of Charlson Comorbidity Index on Return to Recreational and Physical Activities | 2 years postoperatively
  Patient comorbidities will be documented by the surgeon using the weighted Charlson Comorbidity Index. An analysis will be conducted to determine if the index score has a deleterious effect on recreational activities or general fitness activities at follow-up.
Assessment of Postoperative Complications on Return to Recreational and Physical Activities | 2 years postoperatively
  All postoperative complications will be documented in the study patient registry with a list related specifically to TKA from the AKS and a second general list that was generated from complications recorded by the Centers for Medicare and Medicaid Services (2015 update). An analysis will be conducted to determine if complications have a deleterious effect on recreational activities or general fitness activities patients return to after surgery.
Assessment of Effect of Preoperative Body Mass Index on Return to Recreational and Physical Activities | 2 years postoperatively
  Patient body mass index will be collected before surgery and will be designated as either obese, over weight, or within normal limits according to WHO classification of obesity. Determination will be made of the effect of BMI on return to recreational or general fitness activities at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Noyes, MD, Principal Investigator — Cincinnati Sportsmedicine and Orthopaedic Center
Locations (1):
- Cincinnati Sportsmedicine and Orthopaedic Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes